CLINICAL TRIAL: NCT03239561
Title: Phase 0 Exploratory Study of [18F]MNI-1020 (Also Known as [18F]JNJ-64326067) as an Imaging Marker for Tau Protein in the Brain of Subjects With Alzheimer's Disease Compared to Healthy Subjects
Brief Title: Evaluation of Tau Protein in the Brain of Participants With Alzheimer's Disease Compared to Healthy Participants
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CR108349; 64326067EDI0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — JNJ-64326067

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]MNI-1020 (Experimental): Participants will receive a single intravenous bolus injection of [18F]MNI-1020 at a dose of not more than 10 millicurie (mCi), with a maximum mass dose of 10 microgram (mcg) and maximum volume of 10 milliliter (mL) at imaging visit.
  Interventions: Drug: [18F]MNI-1020

INTERVENTIONS:
Drug: [18F]MNI-1020 — Participants will receive a single intravenous bolus injection of [18F]MNI-1020 at a dose of not more than 10 millicurie (mCi), with a maximum mass dose of 10 microgram (mcg) and maximum volume of 10 milliliter (mL) at imaging visit.
  Other Names: [18F]JNJ-64326067

SUMMARY:
The primary objectives of this study are to characterize [18F]molecular neuroimaging (MNI)-1020, a positron emission tomography (PET) radioligand for imaging tau pathology, to visually and quantitatively assess and compare brain uptake and pharmacokinetics of [18F]MNI-1020 in participants with probable Alzheimer's disease (AD) and compare with age matched healthy participants, to evaluate the safety of a single injection of [18F]MNI-1020 and to compare the distribution of tau (using [18F]MNI-1020) and amyloid beta (using florbetapir) in participants with probable AD.

ELIGIBILITY:
Inclusion Criteria:

All Participants

* Female participants must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year. Male participants and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method for male participants for the study duration
* Male participants must not donate sperm during the study and for 3 months after completion

Healthy Participants

* Males and females aged greater than or equal 50 years. Healthy with no clinically relevant finding on physical examination at screening and upon reporting for the [18F]molecular neuroimaging (MNI)-1020 imaging visit
* Have screening [18F]florbetapir positron emission tomography (PET) imaging demonstrating no significant amyloid binding based on qualitative analysis (visual read)

Alzheimer Disease - Have screening [18F]florbetapir or prior amyloid (in the last 12 months) PET imaging demonstrating amyloid binding based on qualitative (visual read)

Exclusion Criteria:

All Participants

* Prior participation in other research protocols or clinical care in the last year in addition to the radiation exposure expected from participation in this clinical study, such that radiation exposure exceeds the effective dose of 50 millisievert (mSv), which would be above the acceptable annual limit established by the United States Federal Guidelines
* Unsuitable veins for repeated venipuncture
* Magnetic resonance imaging exclusion criteria include: evidence of cerebrovascular disease (more than two lacunar infarcts, any territorial infarct greater than 1 centimeter 3, or deep white matter abnormality corresponding to an overall Fazekas scale of 3 with at least one confluent hyperintense lesion on the FLAIR sequence that is greater than or equal to 20 millimeter (mm) in any dimension), infectious disease, space-occupying lesions, normal pressure hydrocephalus or any other abnormalities associated with central nervous system disease
* Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, central nervous system aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in Magnetic Resonance Imaging (MRI)

Alzheimer Disease

- Has received treatment that targeted amyloid beta or tau within the last 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Standardized Uptake Value Ratio (SUVR) of [18F]MNI-1020 | Up to 180 minutes after tracer injection on Day 1
  Tracer uptake will be expressed in Standardized Uptake Value Ratio (SUVR). Regions used for tracer uptake quantitation will include cortical regions (frontal cortex, posterior cingulate, lateral temporal cortex, parietal cortex, occipital cortex, mesial temporal cortex, inferior temporal cortex, hippocampus, and anterior cingulate). Subcortical regions (basal ganglia, substantia nigra, choroid plexus) will be used for detection of possible off-target binding. Regions predicted to be free of tau pathology will be used as reference (cerebellum and pons). SUVR will be calculated as SUV target/SUV reference region (e.g., cerebellar gray).
Plasma Concentration of 18F]MNI-1020 in AD Participants Compared With age Matched Healthy Participants | Pre-injection, 5, 10, 30, and 60 minutes post-injection
  Pharmacokinetics of [18F]MNI-1020 will be assessed by using plasma concentration data and compared in participants with probable Alzheimer's disease (AD) and age matched healthy participants.
Number of Participants With Adverse Events | Baseline up to Follow-Up (Day 4)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Distribution of tau (Using [18F]MNI-1020) Compared to Amyloid Beta (Using Florbetapir) in Participants With Probable AD | Screening for Florbetapir; Day 1 for [18F]MNI-1020
  Within the AD participants, the distribution and binding of [18F]florbetapir will be compared to the [18F]MNI-1020 binding across multiple regions. This will be done by visual reading of scans, with amyloid signal predicted to be high in frontal cortical regions in participants with probable AD and absent from cortex in healthy participants, while tau signal is predicted to be present in hippocampus and entorhinal cortex in healthy elderly participants, and in medial and lateral temporal cortex in participants with probable AD. Semi-quantitative analysis will also be conducted comparing SUVR of the tracers in these same regions, using cerebellum as reference.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Invicro, New Haven, Connecticut, United States